CLINICAL TRIAL: NCT01141673
Title: Development of a Diagnostic Kit for FLT3-ITD in Acute Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Hsingjin Eugene Liu, MD PhD, Taipei Medical University WanFang Hospital
Other Study IDs: FLT3-ITD KIT
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: FLT3-ITD; acute myeloid leukemia; FLT3; D835
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
FLT3 overexpression in acute myeloid leukemia (AML) is often caused by mutations in this gene. These mutations cause constitutive phosphorylation of FLT3 proteins leading to increased proliferation and survival, decreased apoptosis and resistance to chemotherapeutic agents in AML cells. There are two major types of FLT3 mutations- internal tandem duplication (ITD) and point mutation at 835th amino residue. AMLs with FLT3 mutations have worse prognosis and are often resistant to conventional chemotherapy. Several small molecule compounds targeting FLT3 have been in the market or in clinical trials. Therefore, identification of these mutations at the time of diagnosis will provide a better prognostic prediction, might guide the treatment selection and follow-up strategies. In this study, the investigators will develop a sensitive molecular assay to detect FLT3 mutations for future clinical application. The investigators will collect 100 AML samples with at least 20 samples with known FLT3 mutations. The investigators will compare this assay with commonly used methods and standardize the procedure to meet the requirement of clinical pathology laboratory with reasonable cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of acute myeloid leukemia

Exclusion Criteria:

* non

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: acute myeloid leukemia patient in wanfang hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-06; Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Gjin Eugene Liu, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan